CLINICAL TRIAL: NCT06412523
Title: Device-related Central Nervous System Infections in Adult Intensive Care Units in Brazil
Acronym: IMPACTO-SNC
Status: Active, not recruiting | Type: Observational
Sponsor: Beneficência Portuguesa de São Paulo (Other)
Responsible Party: Principal Investigator, Viviane Cordeiro Veiga, MD, PhD, Principal Investigator, Beneficência Portuguesa de São Paulo
Other Study IDs: 17558
Record Dates: First submitted 2022-08-11; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Central Nervous System Infections
Keywords: Central Nervous System Infections; Catheters
MeSH Terms: conditions — Central Nervous System Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Resistant microorganisms are public health problems because they affect the treatment of infectious diseases and the survival of patients. Neurosurgical procedures with placement of intracranial pressure monitoring and external ventricular drainage devices are related to increased morbidity and mortality. In Brazil, there are several multicenter studies demonstrating the prevalence and types of resistant microorganisms, however, there is a lack of data related to central nervous system infections associated with invasive devices, which can have a direct impact on prevention and treatment policies.

DETAILED DESCRIPTION:
Neurosurgical procedures with placement of devices are related to increased morbidity and mortality. A study shows that the incidence of device-related central nervous system infection can reach 27%. A meta-analysis published in 2015, which included 35 studies, showed an incidence of 11.4 per 1000 catheters-day.

This is a prospective cohort study, including adult patients, in the ICUs of hospitals participating in the IMPACTO MR Platform, who have a catheter device for monitoring intracranial pressure or external ventricular shunt, with infection densities and microbiological profile being evaluated; risk factors; clinical management; costs involved and short- and long-term clinical outcomes

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years of age admitted to the ICU in the selected hospitals during the study period, using intracranial pressure monitoring catheters and/or external ventricular shunt.

Exclusion Criteria:

* Diagnosis of brain death.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults admitted to Intensive Care Units.
Sampling Method: Probability Sample
Enrollment: 554 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence density of central nervous system infection | 30 days after study inclusion
  Incidence density will be reported as number of CNS infections per 1000 catheters/day, together with 95% CI. Cumulative incidence will also be reported.

SECONDARY OUTCOMES:
Microbiological characteristics | 30 days after study inclusion
  Microbiological characteristics of device-related central nervous system infections, considering the prevalence of microorganisms (multi-resistant or not)
Risk factors | 30 days after study inclusion
  Risk factors for the development of central nervous system infections in the population studied: institution-associated, operator-associated, patient-associated
Treatment | 30 days after study inclusion
  Treatment practices, focusing on: antimicrobials (time and duration) and focus management (device removal versus maintenance)
Costs | 30 days after study inclusion
  Costs associated with the duration of infection
Deaths | 30 days and 6 months after study inclusion
  Deaths during hospital stay and long-term (6 months)
Rankin scale | 30 days and 6 months after study inclusion
  Measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.
  The patient is classified as follows:
  * No symptoms at all;
  * No significant disability despite symptoms; able to carry out all usual duties and activities
  * Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  * Moderate disability; requiring some help, but able to walk without assistance
  * Moderately severe disability; unable to walk and attend to bodily needs without assistance
  * Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  * Dead

CONTACTS AND LOCATIONS:
Overall Officials: Viviane Veiga, PhD, Principal Investigator — Beneficencia Portuguesa Sao Paulo
Locations (18):
- Brazil (18):
  - Unimed Vitória, Vitória, Espírito Santo
  - Hospital Geral Cleriston Andrade, Feira de Santana, Estado de Bahia
  - Hospital da Cidade, Salvador, Estado de Bahia
  - Santa Casa de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Santa Casa de Misericórdia de Passos, Passos, Minas Gerais
  - Santa Casa de Misericórdia de São João del Rei, São João del Rei, Minas Gerais
  - Instituto Estadual do Cérebro Paulo Niemeyer (Pró Saúde- Associação Beneficente de Assistência Social e Hospitalar), Rio de Janeiro, Rio de Janeiro
  - Hospital Universitário Onofre Lopes, Natal, Rio Grande do Norte
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Instituto Baía Sul de Ensino e Pesquisa Irineu May Brodbeck, Florianópolis, Santa Catarina
  - Hospital de Amor (Fundação PIO XII - Barretos), Barretos, São Paulo
  - Hospital Unimed Limeira, Limeira, São Paulo
  - Hospital das Clínicas - FMUSP Ribeirão Preto, Ribeirão Preto, São Paulo
  - Hospital e Maternidade Brasil (Rede D´or São Luis), Santo André, São Paulo
  - Beneficência Portuguesa de São Paulo, São Paulo, São Paulo
  - Hospital do Coração, São Paulo, São Paulo
  - Hospital São Luiz Itaim, São Paulo, São Paulo
  - Hospital São Paulo, São Paulo, São Paulo